CLINICAL TRIAL: NCT01939340
Title: Prevalence and Impact of Cachexia in Cancer Patients Undergoing Chemotherapy
Brief Title: Prevalence of Cachexia in Patients Undergoing Chemotherapy
Status: Completed | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Nicole Stobaeus, MSc, Charite University, Berlin, Germany
Other Study IDs: EA4/051/10
Record Dates: First submitted 2013-09-06; First posted 2013-09-11 (Estimated); Last update posted 2013-09-12 (Estimated); Status verified 2013-09

CONDITIONS: Cancer; Cachexia
MeSH Terms: conditions — Neoplasms; Cachexia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Cachexia and low nutritional intake are a common phenomena in cancer patients undergoing chemotherapy. The purpose of this study is to assess prevalence of cachexia and low nutritional intake and the impact on quality of life, fatigue and mortality in patients undergoing chemotherapy. Furthermore interactions between these parameters, tumor disease and chemotherapy, respectively.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing chemotherapy at least in the second cycle.
* Patients who have signed a written Informed Consent.

Exclusion Criteria:

* Patients with implanted pacemaker or defibrillator.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be selected in primary care clinics.
Sampling Method: Probability Sample
Enrollment: 285 (Actual)
Dates: Start 2010-04; Primary Completion 2012-09 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Nutritional intake | 1 day
  Nutritional intake will be assessed by 24h-recall, which will be analysed with regard to macronutritients

SECONDARY OUTCOMES:
Cachexia | 1 day
  Cachexia will be evaluated using the patient-generated Subjective Global Assessment.
Quality of life and fatigue | 1 day
  EORTC QLQ C-30 will be used to assess quality of life and additionally cancer-related fatigue will be evaluated using Brief Fatigue Inventory.
Mortality | 6 months
  Mortality will be assesses via telephone or consultation of the local death register

CONTACTS AND LOCATIONS:
Overall Officials: Jörg-Dieter Schulzke, Prof. Dr., Principal Investigator — Charite University, Berlin, Germany
Locations (1):
- Dept. of Gastroenterology, Infectiology and Rheumatology (including workspace nutrition medicine), Charité Universitätsmedizin Berlin, Berlin, State of Berlin, Germany